CLINICAL TRIAL: NCT03159923
Title: Cardiac Remodeling and Prognosis in Secondar Tricuspid Regurgitation
Acronym: TRAP
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC16_8919_TRAP
Record Dates: First submitted 2017-05-15; First posted 2017-05-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2018-09

CONDITIONS: Remodeling, Cardiac; Tricuspid Regurgitation
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Moderate to severe tricuspid regurgitation (≥ 2/4) diagnosed with echocardiography in patients stabilized. — Moderate to severe tricuspid regurgitation (≥ 2/4) diagnosed with echocardiography in patients stabilized.

SUMMARY:
The aim of this study is to improve the definition of the two main types of secondary tricuspid regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Any patients ≥ 18 years old, with moderate to severe tricuspid regurgitation (≥ 2/4), agreeing to participate ;
* The patients included can be ambulatory patients or stabilized hospitalised patients (meaning patient clinicaly stable, not decompensated, and whose normovolemia has been checked).
* Non opposition of the patient

Exclusion Criteria:

* Patient whose accoustic window is judged by the operator as incompatible with a precise evaluation of the tricuspid regurgitation or anatomy of the right cavity ;
* TR < grade 2 ;
* TR secondary to primary pulmonary hypertension or congenital cardiopathy ;
* Primary tricuspid regurgitation (due to rheumatic heart disease, medication - included benfluorex, due to endocarditis, valvular prolapse, carcinoid syndrom or a cardiac stimulation lead …) ;
* Significant left heart valvulopathy (Mitral regurgitation > grade 2, Aortic insufficiency > grade 2, Mitral stenosis < 2 cm², Aortic stenosis < 1.5 cm²). A valvulopathy sucessfully operated isn't considered as an exclusion criteria;
* Cardiopathy with significative systolic dysfunction (FE< 40%) ;
* Patients whose life expectantcy is less than 1 year due to a pathology independent of the TR (neoplasic process for example) ;
* Patient under judicial protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with moderate to severe tricuspid regurgitation (≥ 2/4) diagnosed with echocardiography, in patients stabilized.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-19 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2023-03-23 (Actual)

PRIMARY OUTCOMES:
Composite criteria : cardiovascular death or unscheduled hospitalizations due to cardiovascular event. | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erwan DONAL, PhD, Principal Investigator — Rennes University Hospital
Locations (17):
- France (17):
  - Chu Amiens-Picardie - Site Sud, Amiens
  - Ap-Hp - Hopital Henri Mondor, Créteil
  - CHU de DIJON - HOPITAL FRANCOIS MITTERAND, Dijon
  - Chu Grenoble - Michallon, Grenoble
  - Ghicl - Hopital Saint Philibert, Lomme
  - Chu Marseille - Hopital Nord, Marseille
  - Hôpital Saint Joseph, Marseille
  - Clinique Du Pont de Chaume, Montauban
  - CLINIQUE du MILLENAIRE, Montpellier
  - Chu de Nancy - Hopital de Brabois, Nancy
  - CHU de NANTES - HOTEL DIEU, Nantes
  - Ap-Hp - Hopital Saint-Antoine, Paris
  - Chu de Bordeaux - Groupe Hospitalier Sud, Pessac
  - CHU de Rennes, Rennes
  - CHU de TOULOUSE - HOPITAL RANGUEIL, Toulouse
  - Clinique NCT+, Tours
  - CHU de TOURS - HOPITAL TROUSSEAU, Tours